CLINICAL TRIAL: NCT05772819
Title: 'Cardiac and Intramuscular Adaptations Following Short-term Exercise Prehabilitation in Unfit Patients Scheduled to Undergo Hepatic- or Pancreatic Surgery'
Acronym: CIRCULATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Nationaal Fonds tegen Kanker (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL83611.042.23
Record Dates: First submitted 2023-02-10; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Prehabilitation; Surgery; Exercise Prehabilitation; Perioperative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging arm (Experimental): Participants are subjected to in-magnet exercise test consisting of in vivo exercise cardiac magnetic resonance (exCMR) imaging and 31P-magnetic resonance spectroscopy (31P-MRS) during exercise testing in a MR-compatible ergometer, before and after the 4-week prehabilitation program.
  Interventions: Diagnostic Test: exercise MRI

INTERVENTIONS:
Diagnostic Test: exercise MRI — All patients are subjected to two types of in-magnet exercise tests consisting of exercise cardiac magnetic resonance imaging (exCMR) and Phosphorus 31 magnetic resonance spectrography (31P MRS) of the quadriceps muscle, during exercise at various exercise intensities in a supine position using a MR-compatible ergometer (Lode MR Ergometer Pedal, Lode BV, Groningen, the Netherlands).

SUMMARY:
Surgery remains an important treatment modality in the treatment of hepatopancreatobiliary (HPB) malignancies, but the physiological stress caused by surgery is at the same time a challenge for the homeostasis of patients. A patient's preoperative aerobic capacity has been found to have a consistent relation with postoperative outcomes in major abdominal surgery, with low aerobic capacity being associated with a higher risk of postoperative morbidity and mortality. Preoperative exercise prehabilitation programs can effectively increase the ability of patients to cope with surgical-induced allostatic load, by improving aerobic capacity, and functioning of the respiratory, cardiovascular, and/or musculoskeletal systems. However, besides the effect of exercise prehabilitation on physical fitness in terms of improvement of aerobic capacity as measured by the cardiopulmonary exercise test (CPET), the exact role of adaptations in cardiac and/or skeletal muscle function contributing to the improvement in aerobic capacity is still unknown. Insight in the physiological adaptations that lead to improvement in aerobic capacity after prehabilitation in patients with low aerobic capacity will enable caregivers to individually optimize the exercise program (e.g. by changing exercise frequency, intensity, duration and type) and better explain the rationale and effectiveness behind the short-term physical exercise training program to patients. Therefore, the main objective of this study is to assess the central (cardiac function) and peripheral (skeletal muscle function) physiological adaptations in response to short-term exercise prehabilitation. Secondary objective is to assess the relationship between immune function and exercise. In this study, unfit patients are asked to undergo additional in-magnet exercise testing to investigate the central and peripheral physiological adaptations in response to exercise prehabilitation.

DETAILED DESCRIPTION:
Rationale: Surgery remains an important treatment modality in the treatment of hepatopancreatobiliary (HPB) malignancies, but the physiological stress caused by surgery is at the same time a challenge for the homeostasis of patients. A patient's preoperative aerobic capacity has been found to have a consistent relation with postoperative outcomes in major abdominal surgery, with low aerobic capacity being associated with a higher risk of postoperative morbidity and mortality. Preoperative exercise prehabilitation programs can effectively increase the ability of patients to cope with surgical-induced allostatic load, by improving aerobic capacity, and functioning of the respiratory, cardiovascular, and/or musculoskeletal systems. However, besides the effect of exercise prehabilitation on physical fitness in terms of improvement of aerobic capacity as measured by the cardiopulmonary exercise test (CPET), the exact role of adaptations in cardiac and/or skeletal muscle function contributing to the improvement in aerobic capacity is still unknown. Insight in the physiological adaptations that lead to improvement in aerobic capacity after prehabilitation in patients with low aerobic capacity will enable caregivers to individually optimize the exercise program (e.g. by changing exercise frequency, intensity, duration and type) and better explain the rationale and effectiveness behind the short-term physical exercise training program to patients.

Objective: The main objective is to assess the central (cardiac function) and peripheral (skeletal muscle function) physiological adaptations in response to short-term exercise prehabilitation. Secondary objective is to assess the relationship between immune function and exercise.

Study design: This study is a single-center prospective clinical trial with a one-group pretest-posttest design. It will take place at the University Medical Center Groningen (UMCG), the Netherlands. As part of standard care, all patients scheduled to undergo hepatic or pancreatic surgery for (suspected) HPB malignancies at the UMCG are screened for low aerobic capacity, and subjected to exercise prehabilitation in case of low aerobic capacity. In this study, unfit patients are asked to undergo additional in-magnet exercise testing to investigate the central and peripheral physiological adaptations in response to exercise prehabilitation.

Study population: Unfit patients diagnosed with a (suspected) HPB malignancy who are scheduled to undergo elective hepatic or pancreatic surgical resection and participate in the exercise prehabilitation program. Intervention: In-magnet exercise test consisting of in vivo exercise cardiac magnetic resonance (exCMR) imaging and 31P-magnetic resonance spectroscopy (31P-MRS) during exercise testing in a MR-compatible ergometer, before and after the 4-week prehabilitation program. In addition to exCMR imaging and 31P-MRS during rest, blood will be withdrawn at three different time points (before first CPET, after first CPET and before second CPET).

Main study parameters/endpoints: The difference in left and right ventricular function will be measured by exCMR in rest, during progressive exercise, and recovery to assess the effect of the preoperative physical exercise training program on cardiac function. The difference in quadriceps phosphocreatine concentration (PCr), quadriceps inorganic phosphorus concentration (Pi), and quadriceps pH at rest, during progressive exercise, and recovery rate will be measured by 31P-MRS to assess the effect of the prehabilitation program on skeletal muscle function. Differences in inflammatory and immunological cytokines and chemokines before the first CPET, directly after the first CPET and before second CPET.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The intervention consists of four extra hospital visits. During these visits the in-magnet exercise tests and blood sample collection (exCMR and 31P-MRS) will be performed. The in-magnet exercise test can lead to physical discomfort, due to an uncomfortable feeling while cycling on an ergometer whilst laying supine in the MRI. However, before the in-magnet exercise test, a CPET in a controlled environment (continuous 12-lead electrocardiography registration and under supervision of a sports physician) is performed and therefore the in-magnet exercise test can be safely performed when the CPET does not show contra-indications for exercise. The imaging consisting of exCMR and 31P-MRS has previously been shown to be safe and is already widely used in different studies at the UMCG. Patients are not exposed to any radiation and/or contrast agents. The blood samples that will be taken are not expected to cause an extra risk/burden to the patients. Except for little pain/discomfort, or the possibility of local hemorrhage which can easily solved by compression of the vein

ELIGIBILITY:
Inclusion Criteria:

* VO2 at the VAT ≤13 ml/kg/min and/or VO2peak ≤18 ml/kg/min, as determined during the baseline CPET;
* More than 18 years of age;
* Scheduled for elective liver- or pancreatic resection at the UMCG;
* Willing to participate in the home-based bimodal prehabilitation program;
* Has given consent to participate in the study.

Exclusion Criteria:

* Patients requiring acute (emergency) surgery;
* Patients not capable of cycling on a cycle ergometer;
* Patients with contraindications to physical exercise training;
* Patients receiving neoadjuvant chemotherapy
* Contraindications for exCMR (e.g., claustrophobia, implanted cardiac devices)
* Atrial fibrillation or other significant arrhythmia during the CPET;
* Body weight >140 kg;
* Body height >190 cm;
* History of myocardial infarction, percutaneous coronary intervention or coronary artery bypass graft <3 months or untreated severe obstructive coronary artery stenosis;
* More than moderate left-sided valve disease;
* Complex congenital heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Central physiological adaptations | through study completion, an average of 1 year
  Central adjustments will be determined by differences in LV/RV diastolic strain rate, LV and RV volumes, slope of early LV/RV filling, left and right atrial reservoir strain and emptying fraction, pulmonary artery distensibility and pulsatility, and cardiac output measurements using exCMR, before and after the prehabilitation program.
Peripheral physiological adaptations | through study completion, an average of 1 year
  Peripheral adjustments will be determined by differences in quadriceps PCr, Pi and pH at rest and during progressive exercise and post-exercise recovery rates of quadriceps PCr, Pi and pH using 31P MRS, before and after the prehabilitation program.

SECONDARY OUTCOMES:
Postoperative outcomes | through study completion, an average of 1 year
  Secondary outcomes are perioperative and postoperative outcomes. Postoperative outcomes include overall postoperative complications within 30 days after surgery, grade of complication according to the Clavien-Dindo classification 36 , length of hospital stay in days after surgery, mortality within 30 days after surgery, and readmissions within 30 days after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wijma AG, Driessens H, Jeneson JAL, Janssen-Heijnen MLG, Willems TP, Klaase JM, Bongers BC. Cardiac and intramuscular adaptations following short-term exercise prehabilitation in unfit patients scheduled to undergo hepatic or pancreatic surgery: study protocol of a multinuclear MRI study. BMJ Open Gastroenterol. 2023 Nov 23;10(1):e001243. doi: 10.1136/bmjgast-2023-001243. PMID 37996121